CLINICAL TRIAL: NCT04016597
Title: Comparison of Two Commercially Available Devices to Measure Nitric Oxide Lung Diffusing Capacity in Healthy, Non-smoking Adults
Brief Title: Nitric Oxide Lung Diffusing Capacity in Healthy, Non-smoking Adults
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00226
Record Dates: First submitted 2019-07-04; First posted 2019-07-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: diffusing capacity; reliability; healthy; adults; nitric oxide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung diffusing capacity measurements: Participants perform single-breath lung diffusing capacity measurements in random order during one study visit.
  Interventions: Device: Jaeger Masterscreen TM; Device: HypAir Medisoft

INTERVENTIONS:
Device: Jaeger Masterscreen TM — Single-breath nitric oxide lung diffusing capacity
Device: HypAir Medisoft — Single-breath nitric oxide lung diffusing capacity

SUMMARY:
The measurement of nitric oxide lung diffusing capacity (DLNO) has been recently standardised. To date, two pulmonary function devices are commercially available and are used for the measurement of DLNO. No previous study assessed differences in gas exchange outcomes (e.g., DLNO values) between both devices.

The aim of this project is to compare two commercially available devices that measure lung diffusing capacity for nitric oxide (DLNO).

1. "MasterScreenTM" (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany
2. "HypAir" ("HA", Medisoft, Dinant, Belgium).

DETAILED DESCRIPTION:
In a single-center, crossover study conducted at the University Hospital Zurich, Switzerland, 35 healthy, non-smoking adults (>=18 years) will be invited to perform DLNO measurements in random order using the MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium) devices during one study visit.

The order of the tests on the MasterscreenTM and HypAir devices will be randomly allocated using central randomisation.

ELIGIBILITY:
Inclusion Criteria:

- Age 18 years and older

Exclusion Criteria:

* Previous thoracic surgery
* Smoking
* Chronic lung disease (e.g., asthma bronchiale, COPD)
* Forced expiratory volume in 1s and/or forced vital capacity below the lower limit of normal based on spirometry [Quanjer et al. Eur Respir J 2005]
* Current respiratory infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy people
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Difference in nitric oxide lung diffusing capacity (mL/min/mmHg) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).

SECONDARY OUTCOMES:
Difference in carbon monoxide lung diffusing capacity (mL/min/mmHg) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in Alveolar volume (L) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in inspiratory volume (L) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in breath-hold time (s) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in inspired concentrations for nitric oxide (in %) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in expired concentrations for nitric oxide (in %) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in inspired concentrations for carbon monoxide (in %) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in expired concentrations for carbon monoxide (in %) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in inspired concentrations for helium (%) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in expired concentrations for helium (%) | 1 day
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in inspired concentrations for oxygen (%) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).
Difference in expired concentrations for oxygen (%) | 1 hour
  Single-breath measurements with MasterScreenTM (PFT Pro, Jaeger, CareFusion, Hoechberg, Germany) and HypAir (Medisoft, Dinant, Belgium).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Radtke, PhD, Principal Investigator — University of Zurich, EBPI, Switzerland
Locations (1):
- University of Zurich and University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zavorsky GS, Hsia CC, Hughes JM, Borland CD, Guenard H, van der Lee I, Steenbruggen I, Naeije R, Cao J, Dinh-Xuan AT. Standardisation and application of the single-breath determination of nitric oxide uptake in the lung. Eur Respir J. 2017 Feb 8;49(2):1600962. doi: 10.1183/13993003.00962-2016. Print 2017 Feb. PMID 28179436